CLINICAL TRIAL: NCT01417143
Title: Phase II Study of TKI258 (Dovitinib) Monotherapy in Patients With Unresectable Adenoid Cystic Carcinoma
Brief Title: Dovitinib in Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yung-Jue Bang, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1012-047-344
Record Dates: First submitted 2011-08-09; First posted 2011-08-16 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: dovitinib
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Dovitinib) (Experimental): TKI258 (Dovitinib): 500 mg daily po medication with 5 days on/2 days off schedule. TKI258 (Dovitinib) will be provided by Norvatis for the study purpose. One cycle consists of 4 weeks
  Interventions: Drug: TKI258 (Dovitinib):

INTERVENTIONS:
Drug: TKI258 (Dovitinib): — TKI258 (Dovitinib): 500 mg daily po medication with 5 days on/2 days off schedule. TKI258 (Dovitinib) will be provided by Norvatis for the study purpose. One cycle consists of 4 weeks

SUMMARY:
The purpose of this phase II study of TKI258 (Dovitinib) in adenoid cystic carcinoma is to evaluate the efficacy of TKI258 (Dovitinib).

DETAILED DESCRIPTION:
open, uncontrolled, multi-center, phase II study

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenoid cystic carcinoma
* Local, locally advanced or metastatic disease documented as having shown progression on a scan (CT, MRI, MIBI scan) taken 2 to 12 months prior to baseline compared to a previous scan taken at any time in the past. Progression must be documented according to RECIST criteria.
* Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent and who is previously treated with chemotherapy or local treatment (e.g. transarterial chemoembolization)
* Presence of at least one measurable target lesion for further evaluation according to RECIST criteria
* 18 years or older
* ECOG performance status 0, 1
* Previous treatment with chemotherapy, targeted agents, loco-regional therapy (e.g. chemoembolization) are permitted providing that toxicity has resolved to < or = grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.
* Adequate organ function
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
* A patient who signed the informed consent prior to the participation of the study and who understands that he or she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* A patient with no measurable disease
* Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry)
* A patient with previous active or passive immunotherapy
* A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
* A pregnant or lactating patient
* A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
* A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
* A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin and cervical carcinoma in situ.
* A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
* A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
* Ongoing cardiac arrhythmia of grade > or = 2, atrial fibrillation of any grade, or QTc interval > 450 msec for males or > 470 msec for female.
* A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs
* A patient with peripheral neuropathy of grade 1 by NCI CTC, caused by other factors (e.g. alcohol, diabetes, etc). If the absence of deep tendon reflexes is the only neurologic disorder, this condition does not apply to the exclusion criteria.
* A patient with organ transplantation requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
progression free survival | 4 month
  To determine 4month progression-free survival of TKI258 (Dovitinib) when administered as monotherapy in patients with unresectable adenoid cystic carcinoma

SECONDARY OUTCOMES:
overall survival | 2 years
response rate | 8 weeks
  CT scan will be evaluated every 2 cycles (per 8 weeks)till progression. Reponse rate will be evaluated by RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Seoul National University Hospital, Seoul, South Korea